CLINICAL TRIAL: NCT02631564
Title: An Observational Study of TACE Hepatic Arterial Infusion of Oxaliplatin, Irinotecan and Raltitrexed Treatment for Refractory Liver Metastasis From Colorectal Cancer
Brief Title: Safety of TACE With Oxaliplatin, Irinotecan and Raltitrexed for Refractory Colorectal Cancer Liver Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Bo Zhou, M.D, Ph.D, Fudan University
Other Study IDs: Ral-1
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Colon Cancer Liver Metastasis
Keywords: mCRC;TACE;hepatic infusion;raltitrexed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to observe whether hepatic infusion by oxaliplatin, irinotecan and raltitrexed with or without embolization by lipiodol or microspheres are effective in the treatment of refratory liver metastasis from colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer is one of most popular cancer worldwide. Patients with liver metastasis have poor prognosis except for curative resection. Chemotherapy combined biologic agents have improved mCRC median progress free survival and median overall surivival, but it is difficult to deal with liver lesions after FOLFOX and FOLFIRI treatments failed. We aim to observe the safety and efficacy of hepatic infusion and embolization of oxaliplatin, irinotecan and raltitrexed treatment for refratory liver metastasis from colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed adenocarcinoma of the colon or rectum that is metastatic to the liver and for which standard curative measures do not exist
* Patients must have received prior irinotecan-based treatment for their disease and had documented progression by RECIST criteria; patients must also have received prior fluoropyrimidine and oxaliplatin-based therapy
* Liver disease must not be amenable to potentially curative surgical resection
* Patients must have liver-only or liver-predominant disease to be eligible for this study; hepatic disease must be dominant, but patients are allowed to have extrahepatic disease provided it is not judged likely to be life threatening within 3 months
* Patients must have a patent portal vein as documented by CT, MRI, or ultrasound
* Prior radiation therapy is allowed but must have been completed >= 4 weeks prior to study entry; patients with history of prior radiation to the liver including radio-labeled microspheres cannot take part in this study
* Eastern Cooperative Oncology Group performance status 0-1
* Previous surgery or RFA to the liver is allowed; patients with history of chemoembolization or radio-labeled microspheres are excluded
* Life expectancy of >= 12 weeks
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< ULN
* AST(SGOT)/ALT(SGPT)/Alkaline Phosphatase =< 2.5 X institutional ULN
* Creatinine < 2.0 mg/dL
* PT/PTT < 1.5 X ULN
* Women of childbearing potential (WOCBP) and sexually active males must agree to use an accepted and effective method of contraception prior to study entry and for the duration of the study; WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal; even women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy) should be considered to be of child bearing potential
* Patients must demonstrate ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Hepatic decompensation, or the presence of hepatic encephalopathy Before entering the study with gastrointestinal bleeding within 30 days
* Pregnant or nursing women may not participate in this trial because of the increased risk of fetal harm including death from the therapeutic agents
* Patients with known brain metastases are excluded from this study because of their poor prognosis and frequent development of progressive neurological dysfunction that would confound the evaluation of neurologic and other adverse events
* As patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, known HIV-positive patients and those with known hepatitis B or C are excluded from the study Uncontrolled intercurrent illness including, but not limited to, ongoing or active bacterial infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with clinically evident ascites requiring medical management or paracentesis, or Childs-Pugh score B/C are not eligible
* Patients with evidence of other cancer within 5 years, excluding adequately treated basal cell carcinoma of the skin
* Patient with significant cardiac, renal or hematologic or pulmonary dysfunction
* Patients with previous chemoembolization to liver metastases Patients may not receive any other anticancer therapy while on study, including immunotherapy; patients may not receive any other clinical investigational drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Refractory liver metastasis from colon and rectal cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
number of adverse events | 6 months

SECONDARY OUTCOMES:
Overall survival | 2 years
Time to progression | one year

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhou, M.D,Ph.D, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided